CLINICAL TRIAL: NCT05288426
Title: Consequences of Post BNT162b2 Vaccine Myocarditis and Multiple Inflammatory Syndrome Myocarditis
Brief Title: Myocarditis Post Vaccination or Multi System Inflammatory Syndrome
Acronym: MyoVax
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Mevorach Dror, Professor & Head, Department of Internal Medicine B; Head, Rheumatology Research Center, Hadassah and the Hebrew University Medical School, Hadassah Medical Organization
Other Study IDs: DM005
Record Dates: First submitted 2021-12-13; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained from patients with post vaccine (BNT162b2 vaccine ) myocarditis, or MIS following a consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- participant post first BNT162b2 vaccination: Patients which developed myocarditis after the first dose of BNT162b2 vaccination
  Interventions: Other: No intervention
- participant post second BNT162b2 vaccination: Patients which developed myocarditis after the second dose of BNT162b2 vaccination
  Interventions: Other: No intervention
- participant post third BNT162b2 vaccination: Patients which developed myocarditis after the third dose of BNT162b2 vaccination diagnosed with MIS
  Interventions: Other: No intervention
- participant post COVID-19: Patients which developed myocarditis after COVID-19 infection
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, with no intervention.

SUMMARY:
BNT162b2 vaccine has become one of the most prevalent vaccines against the COVID-19 and is currently the main vaccine used in Israel. Since marketing and the beginning of use of the vaccine, we and others have reported. of the development of post vaccination myocarditis.

In this study the investigators wish to explore the long term impact on 150 patients who have been diagnosed with myocarditis or multisystem inflammatory syndrome (MIS) in the year following their diagnosis of Myocarditis.

DETAILED DESCRIPTION:
Aim of Study

The primary aim of the study is to evaluate the impact of long term impact of myocarditis which has been developed secondary to Covid 19 vaccine or Covid 19 infection.

The primary end points of the study will be functional evaluations of the patients using clinical evaluation that includes questionnaires, ECG findings, evaluation of the systolic and diastolic function of the heart using echocardiogram or cardiac MRI, laboratory tests including troponin, CPK, CRP, Pro-BNP, and cytokines/chemokines.

Methods In this prospective study patients will be recruited from health care providers The selected patients will come to Hadassah hospital within 6 and 12 months after they have been diagnosed with myocarditis. Upon the patients arrival they will sign the informed consent, the investigators will draw blood tests and the participants will perform an echocardiogram according to the special protocol and will perform cardiac- MRI according to the myocarditis protocol. Patients will fulfill health questionnaires. that may include 36 Health Survey Questionnaire (SF-36); Scores on the European Quality of Life-5 Dimensions (EQ-5D) survey, which is also health-related quality of life score; the Scores on the European Quality of Life Visual Analogue Scale (EQ-VAS); Kansas City Cardiomyopathy Questionnaire (KCCQ). the Investigators will obtain blood samples from all the patients: complete blood count, c- reactive protein, troponin, CPK, Pro-BNP, liver and kidney functions, magnesium and cytokines. In addition, all participants will undergo echocardiogram test to evaluate their systolic and diastolic function of the heart.

Ethical Considerations

The study poses no danger to the participants. It has the potential to improve the understanding of the impact myocarditis post COVID-19 MRNA vaccine on the quality of life of those patients and provide a descent follow-up for the participant. Any participant will sign on informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females.
* Minors male and female.

Diagnosed as myocarditis:

* Evidence of myocarditis on biopsy or increased biomarkers of myocardial injury (TNI and CK-MB and BNP or NT-pro-BNP)
* Acute onset of symptoms of cardiac dysfunction: dyspnea, palpation, chest pain, and/or syncope;
* Image for cardiac injury: marked diffused reduction in left ventricle wall movement, with dramatically decreased left ventricle ejection fraction (LVEF) < 45%, or by cardiac magnetic resonance imaging.

Exclusion Criteria:

* Also considering acute coronary syndrome but unable to perform coronary angiography to distinguish acute coronary syndrome from myocarditis, or otherwise suffer from valvuloplasty.
* Myocardial injury caused by sepsis, medical agents, or poisons;
* Malignancy or any comorbidity limiting survival or conditions predicting inability to complete the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were hospitalized at Hadassah Medical Center and other hospitals in Israel, with the diagnosis of myocarditis post COVID-19 or post BNT162b2 vaccine (as specified in the inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess troponin levels in patients that developed acute myocarditis | 3 years
  troponin levels in each clinical visit will be documented
To assess PRO-BNP levels in patients that developed acute myocarditis | 3 years
  PRO-BNP levels in each clinical visit will be documented
To assess CRP levels in patients that developed acute myocarditis | 3 years
  CRP levels in each clinical visit will be documented
To assess cardiac MRI in patients that developed acute myocarditis | 3 years
  Cardiac MRI will be performed at least yearly and evaluated for regionally increased signal in T2-weighted images; Late gadolinium enhancement in a nonischemic pattern, Increased native T1 values on a 3T magnet.
To assess echocardiogram in patients that developed acute myocarditis | 3 years
  echocardiogram will be performed at least yearly and defined as normal, ST-segment elevation, with Diffuse or Non-diffuse changes, T-wave changes, Atrial fibrillation or non-sustained ventricular tachycardia.
To assess health quality by a questionnaire in patients that developed acute myocarditis | 3 years
  EQ-5D will be fill at least once a year. Descriptive analysis of EQ-5D profile at each observation and analysis of changes between repeated observations. Cluster analysis can be used.
To assess heart failure questionnaire in patients that developed acute myocarditis | 3 years
  KCCQ will be fill at least once a year.

SECONDARY OUTCOMES:
Cytokine in Patients after myocarditis | 3 years
  To assess cytokines by measuring the serum concentrations
Chemokine in Patients after myocarditis | 3 years
  To assess chemokines by measuring the serum concentrations
Hematopoietic Growth Factors (HGF)in patients after myocarditis | 3 years
  To assess Hematopoietic Growth Factors in patients with COVID-19 by measuring the To assess HGF by measuring the serum concentrations
Complement in patients after myocarditis | 3 years
  assess complement factors by measuring the serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mevorach D, Anis E, Cedar N, Bromberg M, Haas EJ, Nadir E, Olsha-Castell S, Arad D, Hasin T, Levi N, Asleh R, Amir O, Meir K, Cohen D, Dichtiar R, Novick D, Hershkovitz Y, Dagan R, Leitersdorf I, Ben-Ami R, Miskin I, Saliba W, Muhsen K, Levi Y, Green MS, Keinan-Boker L, Alroy-Preis S. Myocarditis after BNT162b2 mRNA Vaccine against Covid-19 in Israel. N Engl J Med. 2021 Dec 2;385(23):2140-2149. doi: 10.1056/NEJMoa2109730. Epub 2021 Oct 6. PMID 34614328
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967